CLINICAL TRIAL: NCT03726866
Title: A Randomized, Open Label, Repeated-dose, Crossover Study to Investigate the Pharmacokinetic Drug Interactions and Safety Among D326, D337 and CKD-828 in Healthy Subjects
Brief Title: A Study to Investigate Drug-Drug Interaction Between D326, D337 and CKD-828 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 186DDI18020
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Dyslipidemias; Hypertension
Keywords: dyslipidemias; hypertension; Drug-Drug interaction
MeSH Terms: conditions — Dyslipidemias; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Sequence 1
  Interventions: Drug: Sequence 1
- Sequence 2 (Experimental): Sequence 2
  Interventions: Drug: Sequence 2
- Sequence 3 (Experimental): Sequence 3
  Interventions: Drug: Sequence 3
- Sequence 4 (Experimental): Sequence 4
  Interventions: Drug: Sequence 4
- Sequence 5 (Experimental): Sequence 5
  Interventions: Drug: Sequence 5
- Sequence 6 (Experimental): Sequence 6
  Interventions: Drug: Sequence 6

INTERVENTIONS:
Drug: Sequence 1 — D326, D337 or CKD-828 for 9 days
  Arms: Sequence 1
Drug: Sequence 2 — D326, D337 or CKD-828 for 9 days
  Arms: Sequence 2
Drug: Sequence 3 — D326, D337 or CKD-828 for 9 days
  Arms: Sequence 3
Drug: Sequence 4 — D326, D337 or CKD-828 for 9 days
  Arms: Sequence 4
Drug: Sequence 5 — D326, D337 or CKD-828 for 9 days
  Arms: Sequence 5
Drug: Sequence 6 — D326, D337 or CKD-828 for 9 days
  Arms: Sequence 6

SUMMARY:
To evaluate pharmacokinetic properties and drug interactions between D326 and D337 co-administered groups, the CKD-828 alone and the total co-administered groups.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged between ≥ 19 and ≤ 40 years old
2. Calculated body mass index(BMI) of ≥ 19 and ≤ 28kg/m²
3. Subject who agree to use a combination of effective contraceptive methods or medically acceptable contraceptive methods from the date of first administration of Investigational product until completion of the clinical trial
4. Subject who agree not to provide sperm
5. Subject who voluntarily agree to participate in this study

Exclusion Criteria:

1. Any medical history that may affect drug absorption, distribution, metabolism and excretion
2. Subject who has a clinically significant disease or history such as endocrine, gastrointestinal, cardiovascular, muscular disease.
3. Genetic problems such as galactose intolerance, Lapp lactose dehydrogenase deficiency or glucose-galactose uptake disorder
4. Subject who have received other clinical trial drugs within 90 days prior to the screening visit
5. Any clinically significant active chronic disease

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-01-15 (Estimated); Study Completion 2019-01-15 (Estimated)

PRIMARY OUTCOMES:
Cmax(Maximum plasma concentration of the drug at steady state) | at Day 9
  PK parameters of D326, D337 and CKD-828
AUCtau(area under the plasma concentration-time curve for a dosing interval at steady state) | at Day 9
  PK parameters of D326, D337 and CKD-828

SECONDARY OUTCOMES:
Tmax(Time to maximum plasma concentration at steady state) | at Day 9
  PK parameters of D326, D337 and CKD-828
t1/2(Terminal elimination half-life) | at Day 9
  PK parameters of D326, D337 and CKD-828

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong-Seok Lim, M.D., Ph.D., Principal Investigator — Department of Clinical Pharmacology and Therapeutics / Asan Medical Center, University of Ulsan
Locations (1):
- Asan Medical Center, University of Ulsan, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No